CLINICAL TRIAL: NCT03246685
Title: A Multicenter, Open-label, Phase 2 Study of Imprime PGG & Pembrolizumab in Subjects With Adv Squamous Cell Carcinoma of H&N (SCCHN) Who Failed Pembro Monotherapy or Experiencing SD Following Completion of 4 to 8 Cycles of Pembro Monotherapy
Brief Title: Phase 2 Study of Imprime PGG & Pembrolizumab in Subjects With Adv SCCHN Who Failed Pembro Monotherapy or Experiencing SD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to enrollment challenges resulting in changing treatment patterns, the study has been terminated. No patients remain on study.
Sponsor: HiberCell, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-CL-PGG-HNC-1622MK3475PN-544
Record Dates: First submitted 2017-07-22; First posted 2017-08-11 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab Failures (Experimental): Imprime PGG + Pembrolizumab
  Interventions: Biological: Imprime PGG; Drug: Pembrolizumab
- Active Stable Disease on Pembrolizumab (Experimental): Imprime PGG + Pembrolizumab
  Interventions: Biological: Imprime PGG; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Imprime PGG — Imprime PGG is a soluble, β-1,3/1,6 glucan isolated from the cell wall of a proprietary Saccharomyces cerevisiae yeast strain. Imprime PGG acts as a Pathogen-Associated Molecular Pattern (PAMP). Imprime will be administered at a dose of 4 mg/kg IV over a 2-hour infusion time on Days 1, 8 and 15 of each 3-week treatment cycle.
  Other Names: Imprime
Drug: Pembrolizumab — Pembrolizumab is a humanized monoclonal antibody against the programmed death receptor-1 protein. Pembrolizumab will be given at a fixed dose of 200 mg IV over 30 minutes on Day 1 of each 3-week treatment cycle after the Imprime infusion.
  Other Names: Keytruda

SUMMARY:
Objective: To determine the Overall Response Rate (ORR) to Imprime PGG + pembrolizumab in subjects with advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN) Safety: To characterize the safety of Imprime PGG + pembrolizumab given in combination Hypothesis: Restore (for subjects who have failed pembrolizumab mono therapy) or enhance (for subjects who actively experiencing SD) sensitivity to checkpoint inhibitors (CPI) by appropriate and effective stimulation of the subject's innate and adaptive immune systems by combining Imprime PGG with pembrolizumab.

The study will require documenting at least 5 objective responses among the 38 subjects enrolled who have failed prior pembrolizumab monotherapy and at least 17 objective responses among the 49 subjects enrolled who are actively experiencing stable disease following at least 4 cycles (but no more than 8 cycles) of pembrolizumab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed an informed document prior to any study-specific procedures or treatment
2. Be ≥ 18 years of age at time of consent
3. Have histologically or cytologically confirmed diagnosis of SCCHN irrespective of PD-L1 status, which is either inoperable and recurrent, or metastatic
4. Up to 3 prior chemotherapy regimens or metastatic disease
5. Have either:

   1. Investigator determined assessment of disease progression after treatment with pembrolizumab monotherapy, OR
   2. Investigator determined assessment of current stable disease following completion of at least 4 cycles but no more than 8 cycles, of pembrolizumab monotherapy
6. Have resolution of all previous treatment-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy (less than or equal to Grade 2) or alopecia. If subject received major surgery or radiation therapy of > 30 Gy, must have recovered from the toxicity and/or complications from the intervention.
7. Have at least one radiologically measurable lesion as per RECIST v1.1 defined as a lesion that is at least 10 mm in longest diameter or lymph node that is at least 15 mm in short axis imaged by CT scan or MRI and obtained by imaging within 28 days prior to start of study treatment. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. Have peripheral blood levels of IgG anti-β-glucan antibody (ABA) of ≥ 20 mcg/mL as determined by an ELISA test within 90 days prior to start of study treatment
9. Be willing to consider providing fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality, for assessment of biomarker status. Repeat samples may be required if adequate tissue is not provided. Newly obtained biopsy specimens are preferred to archived samples and formalin-fixed, paraffin-embedded block specimens are preferred to slides.

   Note: Information on 1 tumor biopsy sample is mandatory and is as follows: (1) To determine eligibility, historical (diagnostic) tumor biopsy official pathology report +/- an archival sample. Additional biopsy samples, preferably obtained from the same localized region, are highly desirable when feasible at the following time points: (2) Sample before the first dose of study treatment, (3) Sample after completion of Cycle 2 but before the start of Cycle 3 dosing, and (4) Sample either at the time of response or at the End of Study Visit (if no response).
10. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (see Appendix 14.3)
11. Have life expectancy of 6 months or greater as determined by the treating physician
12. Have adequate organ function (all screening labs should be performed within 15 days prior to study treatment):

    1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
    2. Aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
    3. Alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
    4. Albumin level ≥3 g/dL
13. Have adequate renal function within 15 days prior to study treatment, defined by the following criteria:

    Creatinine ≤ 1.5 x ULN and CrCl ≥ 30 ml/min per Cockcroft Gault formula:
14. Have adequate hematologic function within 15 days prior to study treatment, defined as meeting all of the following criteria:

    1. Hemoglobin ≥ 9 g/dL (uncorrected by RBC transfusion)
    2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
    3. Platelet count ≥ 100 × 109/L
15. Have adequate coagulation functioning within 15 days prior to start of study treatment, defined by either of the following criteria:

    1. INR < 1.5 × ULN
    2. OR for subjects receiving warfarin or low molecular weight heparin (LMWH), the subjects must, in the Investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these subjects may exceed 1.5 × ULN if that is the goal of anticoagulant therapy.
    3. Activated Partial Thromboplastin Time (aPTT) < 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
16. Female subjects of childbearing potential as defined in Section 5.7.2 must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
17. If of childbearing potential as defined in Section 5.7.2, must be willing to use an adequate method of contraception (see Section 5.7.2) from the first dose of study medication through 120 days after the last dose of study medication
18. Be willing and have the ability to comply with scheduled visits (including geographical proximity), treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Has disease that is suitable for local therapy administered with curative intent
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
3. Has a diagnosis of immunodeficiency or receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
4. Has known history of active tuberculosis
5. Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
6. Has known active Hepatitis B (eg, HBsAg reactive) or Hepatitis C (eg, HCV RNA [qualitative] is detected
7. Has a history of clinically severe autoimmune disease, or history of organ transplant
8. Has known hypersensitivity to baker's yeast
9. Had previous exposure to Betafectin® or Imprime PGG
10. Has severe hypersensitivity to pembrolizumab or any of its excipients
11. Had a prior anti-cancer monoclonal antibody (other than pembrolizumab) within 30 days prior to start of study treatment, or failure to recover to CTCAE Grade 1 or better from the adverse events of prior therapies
12. Had within 2 weeks prior to the first dose of study treatment, received prior chemotherapy, targeted small molecule therapy, or radiation therapy, or who has not recovered from adverse events due to a previously administered agent or major surgery
13. Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF, or recombinant erythropoietin) within 4 weeks prior to the first dose of study treatment
14. Has known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
15. Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
16. Has active autoimmune disease requiring systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteriod replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
17. Has history of (non-infectious) pneumonitis that required steroids or current pneumonitis
18. Has a history of interstitial lung disease
19. Has an active infection requiring systemic therapy
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator
21. Has a clinically significant cardiovascular disease such as unstable angina, myocardial infarction, or acute coronary syndrome within ≤180 days prior to start of study treatment, symptomatic or uncontrolled arrhythmia, congestive heart failure, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
22. Has a known psychiatric or substance abuse disorder(s) that would interfere with informed consent or cooperation with the requirements of the trial
23. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
24. Has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) to Imprime PGG + pembrolizumab using RECIST v1.1 criteria | Within 18 months of last patient enrolled

SECONDARY OUTCOMES:
Time to response (TTR) using RECIST v1.1 criteria | Within 24 months of last patient enrolled
Complete response rate (CRR) using RECIST v1.1 criteria | Within 24 months of last patient enrolled
Duration of overall response (DoR) using RECIST v1.1 criteria | Within 24 months of last patient enrolled
Progression-Free Survival (PFS) and PFS rate at 6 months and 1 year using RECIST v1.1 criteria | 6 months and 1 year after first dose and within 24 months of last patient enrolled
Overall survival (OS) and OS rate at 1 year | 1 year after first dose and within 24 months of last patient enrolled
Pharmacokinetic (PK) concentration for Imprime PGG and Pembrolizumab | Within 24 months of last patient enrolled

OTHER OUTCOMES:
ORR based on irRECIST | Within 24 months of last patient enrolled
PFS based on irRECIST | Within 24 months of last patient enrolled
Correlate levels of baseline serum anti-β-glucan antibody (ABA) with objective response and treatment outcomes | Within 24 months of last patient enrolled
Correlate changes in immune cell activation markers, such as CD86 expression in tumor biopsy samples and in peripheral blood immune cells with objective response and treatment outcome | Within 24 months of last patient enrolled
In tumor biopsies, correlate changes in the tumor immune microenvironment including TILs (Tumor-infiltrating Lymphocytes) and tumor-infiltrating myeloid cells with objective response and treatment outcome | Within 24 months of last patient enrolled
Correlate PD-L1 expression in tumor biopsy samples (in tumor cells and myeloid cells) with objective response and treatment outcome | Within 24 months of last patient enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medical Specialties, PLLC, Tacoma, Washington, United States